CLINICAL TRIAL: NCT01128309
Title: Stress Reduction and Anxiety: Effects on the Function and Structure of the Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Britta Holzel, Research Fellow, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010P000947; 236975 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress Reduction Intervention (Experimental): Stress Reduction Intervention
  Interventions: Behavioral: Stress Reduction Intervention
- Active Control Condition (Active Comparator)
  Interventions: Behavioral: Active Control intervention

INTERVENTIONS:
Behavioral: Stress Reduction Intervention — eight week group program, plus daily homework practice
  Arms: Stress Reduction Intervention
Behavioral: Active Control intervention — weekly group meetings for eight weeks, plus daily homework practice
  Arms: Active Control Condition

SUMMARY:
The aim of the study is to test whether Generalized Anxiety Disorder (GAD) patients that participate in a Stress Reduction Intervention show a brain activation pattern (assessed by MRI) indicative of improved emotion regulation compared to an active control intervention.

ELIGIBILITY:
Inclusion Criteria:

* participation in the study 'Stress Reduction Techniques and Anxiety: Therapeutic and Neuroendocrine Effects" by Dr. Elizabeth Hoge

Exclusion Criteria:

* metallic implants
* left handed
* epileptic seizures
* head trauma
* weight over 350 pounds
* claustrophobia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
brain activation and structure as assessed by MRI | Day 1 (within two weeks before the intervention)
  BOLD functional MRI and structural MRI
brain activation and structure as assessed by MRI | Day 2 (within two weeks after the intervention)
  BOLD functional MRI and structural MRI

CONTACTS AND LOCATIONS:
Overall Officials: Sara W Lazar, PhD, Principal Investigator — Massachusetts General Hospital; Britta K Holzel, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States